CLINICAL TRIAL: NCT06508645
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-dose Clinical Trial to Evaluate the Safety/Tolerability and Pharmacokinetics, and Pharmacodynamics After Intravenous DWP14012 Injection in Healthy Volunteers
Brief Title: Study to Evaluate the Safety/Tolerability, PK and PD After Intravenous DWJ1521 Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1521102
Record Dates: First submitted 2021-12-15; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — fexuprazan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part1 Treatment Group_1 (Placebo Comparator): Part1 Treatment Group_1_low dose DWP14012 injection Amg, Multiple administration, 7 days
  Placebo: Normal saline
  Interventions: Drug: DWP14012 injection
- Part1 Treatment Group_2 (Placebo Comparator): Part1 Treatment Group_2_medium dose DWP14012 injection Bmg, Multiple administration, 7 days
  Placebo: Normal saline
  Interventions: Drug: DWP14012 injection
- Part1 Treatment Group_3 (Placebo Comparator): Part1 Treatment Group_3_high dose DWP14012 injection Cmg, Multiple administration, 7 days
  Placebo: Normal saline
  Interventions: Drug: DWP14012 injection
- Part2 Treatment Group (Experimental): Part2 Treatment Group_continuous intravenous administration
  - DWP14012 injection Dmg, Loading dose / DWP14012 injection Emg for 3 days, Maintenance dose
  Interventions: Drug: DWP14012 injection

INTERVENTIONS:
Drug: DWP14012 injection — 1. Part 1
     * Study drug: Daewoong Pharmaceutical Co., Ltd.; A mg, B mg, and C mg of DWP14012 inj. (40 mg/vial)
     * Control drug: Placebo (Normal saline)
  2. Part 2 • Study drug: Daewoong Pharmaceutical Co., Ltd.; DWP14012 inj. (40 mg/vial)
  Other Names: Fexuprazan

SUMMARY:
A randomized, double-blind, placebo-controlled, multiple-dose clinical trial to evaluate the safety/tolerability and pharmacokinetics, and pharmacodynamics after intravenous DWP14012 injection in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged ≥ 19 and ≤ 50 years at screening
2. Subjects with a body weight of ≥ 55.0 kg to ≤ 90.0 kg with a body mass index (BMI) of ≥ 18.0 and ≤ 28.0 at screening

   ☞ BMI(kg/m2) = weight (kg) / {Height (m)}2
3. Subjects who have given written consent on voluntary decision of participation prior to the screening procedure after being fully informed of and completely understanding this study
4. Subjects eligible to participate in the study at the discretion of the investigator by physical examination, laboratory tests, investigator questioning, etc.

Exclusion Criteria:

1. Present or prior history of clinically significant hepatic, renal, nervous system, immune, respiratory, and endocrine diseases, hematologic and oncologic diseases, cardiovascular diseases, or mental diseases
2. Gastrointestinal diseases (gastric ulcer, gastritis, gastric cramps, gastroesophageal reflux, Crohn's disease, etc.) that may affect the safety and pharmacokinetic evaluation results of investigational drugs and those with a history of gastrointestinal surgery (except for appendix surgery and hernia surgery alone).
3. Helicobacter pylori positive.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
AUC0-24h of Fexuprazan | Part1 for 8 days, Part2 for 5 days
  Pharmacokinetics parameter following DWP14012 injection
24h pH monitoring, the ratio of the time remaining above pH 4, 6 (time%) | Part1 for 8 days, Part2 for 4 days
  Parmacodynamics parameter following DWP14012 injection

CONTACTS AND LOCATIONS:
Overall Officials: Injin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul-National University Hospital, Seoul, South Korea